CLINICAL TRIAL: NCT00704834
Title: Gene Expression Profiles in Patients With Multiple Sclerosis
Brief Title: Gene Expression Profiles in Multiple Sclerosis (MS)
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 291796
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Relapsing Remitting Multiple Sclerosis; Chronic Progressive Multiple Sclerosis; Clinically Isolated Syndrome; Normal Controls; Blood Draw
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 35cc of peripheral blood will be obtained from each subject via venipuncture.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: Normal Controls
  Interventions: Other: Blood Draw
- 2: Patients with a clinically isolated syndrome (CIS)
  Interventions: Other: Blood Draw
- 3: Patients with relapsing, remitting Multiple Sclerosis (RRMS) who are not on treatment
  Interventions: Other: Blood Draw
- 4: Patients with Chronic Progressive Multiple Sclerosis who are not on treatment
  Interventions: Other: Blood Draw

INTERVENTIONS:
Other: Blood Draw — 35 cc of peripheral blood will be obtained by venipuncture from each subject.

SUMMARY:
The purpose of this study is to test differences in RNA levels between Multiple Sclerosis (MS) patients and normal subjects. RNA provides a "message" from genes altered in diseases. We will also test DNA to determine if there are any small mutations called SNPs in any of the genes. The last tests are two separate tests for markers of inflammation called cytokines and eicosanoids. This research may lead to the discovery of biological markers for MS that are useful for diagnosis and treatment.

DETAILED DESCRIPTION:
This is an investigator-initiated, pilot study of gene expression (RNA) in the blood of patients with multiple sclerosis (MS). The study will enroll patients from the UC Davis Multiple Sclerosis clinic. At a single study visit, we will confirm eligibility, obtain clinical information, and collect blood samples. We will then process these samples to obtain RNA for subsequent microarray analysis. DNA will also be used to examine single nucleotide polymorphisms (SNPs) on chips that allow us to examine 1 million of these SNPs. The SNPs may allow us to diagnose a disease like multiple sclerosis or to predict a treatment or cause. In addition, the DNA may be used to determine if there are any small mutations in any of the genes in the individuals who donate their blood. Additional studies will be done on blood plasma, testing for inflammatory molecules called eicosanoids and cytokines. The data from these tests will be superimposed on the microarray data to determine a molecular profile for each patient. We will then compare the data obtained between patient groups to determine gene alterations specific for each condition.

ELIGIBILITY:
Inclusion Criteria:

* males and females
* any race
* Between the ages of 18 and 70 years
* Diagnosed with a clinically isolated syndrome or the diagnosis of multiple sclerosis using the widely established Macdonald criteria. A 'clinically isolated syndrome' refers to an isolated attack of optic neuritis, transverse myelitis, or brain demyelination. Relapsing-remitting MS is characterized by acute relapses that are followed by some degree of recovery without worsening of disability between relapses. Chronic progressive MS is defined as sustained progression of physical disability, occurring separately from relapses, in patients with MS.
* Control subjects will be male or female, between the ages 18 to 70 years, of any race, with no symptoms of MS.

Exclusion Criteria:

* Children are excluded from the study because MS is generally a disease of young adult onset and is rare in children.
* Evidence of infection or communicable disease, cancer or other known systemic disease, anti-coagulation, known bleeding disorder, illicit drug abuse, or change in medications in the last 30 days (including treatment with steroids).
* Patients receiving any other immune modulating medications (steroids, cyclophosphamide, mitoxantrone, methotrexate, mycophenolate mofetil, azathioprine, IVIG or rituximab) in the prior thirty days will be excluded from the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult subjects aged 18 to 70 will be enrolled. There will be four study groups: patients with a clinically isolated syndrome (CIS), patients with untreated relapsing-remitting MS (RR-MS), patients with chronic, progressive MS (CPMS), and age- and gender-matched control subjects without MS. Patients of both sexes and all races will be recruited into the study without bias.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2006-03; Primary Completion 2017-07-05 (Actual); Study Completion 2017-07-05 (Actual)

PRIMARY OUTCOMES:
Determine MS-specific peripheral blood gene expression patterns | 3 years
Determine differences in peripheral blood gene expression patterns between subgroups of MS patients | 3 years
Determine whether there are specific SNPs correlated with altered gene expression profiles in multiple sclerosis | 3 years
Determine MS-specific peripheral blood inflammatory marker profiles | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Apperson, MD, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No